CLINICAL TRIAL: NCT07009340
Title: Retrospective Observational Study of Patients Who Have Undergone Coronary Artery Bypass Graft (CABG) and/or Cardiac Valve Surgery: Post-discharge Follow-up of Patients From REN-004 Clinical Trial
Brief Title: Retrospective Observational Study of Patients Who Have Undergone Coronary Artery Bypass Graft (CABG) and/or Cardiac Valve Surgery
Status: Active, not recruiting | Type: Observational
Sponsor: Renibus Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: RT-RBT1-RWE01
Record Dates: First submitted 2025-05-29; First posted 2025-06-06 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Post-discharge Outcomes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

SUMMARY:
This study is a retrospective chart abstraction for subjects who were enrolled in REN-004. As a retrospective study, all data will be abstracted from the medical records.

ELIGIBILITY:
Inclusion Criteria:

* Patient completed REN-004
* Patient has at least 1 year of follow documentation post-discharge

Exclusion Criteria:

* Patient enrolled in a clinical trial within 1-year post-discharge from REN-004

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who completed REN-004 and have at least 1 year of follow documentation post-discharge
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-11-18 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Post-discharge outcomes for patients enrolled in REN-004 from one study center | 1 year
  Readmission for any reason Rehospitalization related to procedure/valve/heart failure Contacts with HCP post discharge (any HCP) PCP (if available) All tests and procedures post discharge Medications Chronic kidney disease (CKD) - new diagnosis Acute kidney injury (AKI) requiring dialysis Chronic Kidney disease (CKD) requiring dialysis Atrial fibrillation - new-onset Myocardial infarction (MI) Non-fatal cardiac arrest Reoperation for coronary artery bypass graft (CABG) Reoperation for valve dysfunction Stroke Death from any cause MACCE Death from any cause, repeat revascularization (CABG or PCI), non-fatal MI, and stroke

SECONDARY OUTCOMES:
Total estimated cost of in hospital and post-discharge | 1 year

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Heart Center Research, LLC, Huntsville, Alabama
  - Lutheran Medical Center, Fort Wayne, Indiana
  - My Michigan Medical Center, Midland, Michigan
  - University of Texas Southwestern Medical Center, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No